CLINICAL TRIAL: NCT00755235
Title: Pilot Trial of Depression Care Management by Electronic Secure Messaging
Brief Title: Feasibility of Depression Care Management by E-mail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R21MH082924 (NIH); R21MH082924 (NIH); DSIR 82-SEDR
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: Depression; Primary care; Effectiveness; Care management
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive depression care management by secure messaging.
  Interventions: Other: Depression care management by secure messaging
- 2 (No Intervention): Participants will receive their usual care, with no additional education or care management services.

INTERVENTIONS:
Other: Depression care management by secure messaging — Participants will receive electronic messages welcoming them and monitoring their antidepressant treatment. Care managers will use monitoring data to aid participants' physicians, coordinate physician follow-ups, facilitate emergency care, and facilitate specialty referrals. Care managers will also provide motivation and education to participants.
  Other Names: online messaging; email
  Arms: 1

SUMMARY:
This study will test whether an electronic system that monitors and sends messages to help people with depression could be feasible, acceptable, and potentially effective as a treatment.

DETAILED DESCRIPTION:
Symptoms of depression, such as persistent sadness, problems sleeping, and inability to feel pleasure, interfere with the daily lives of more than 20 million Americans. Previous research indicates that telephone care management systems improve the quality and outcomes of depression care, but are too expensive to be used widely. Using secure messaging over e-mail would be more cost effective than telephone care. This study will examine whether a secure messaging care management program would be feasible, based on whether participants are willing to sign up for and continue with the program, and whether the program has a positive effect on those participants enrolled in the program.

Potential participants for this study will be contacted via e-mail, with a follow-up telephone call if they do not respond to the e-mail message. Only people who have used e-mails in the past year and who are starting antidepressant treatment will be contacted. The percentage of people contacted who enroll will be recorded.

Participation in this study will last 6 months. Participants will be randomly assigned to receive either a secure messaging care management program, based on effective telephone management programs, or their usual care with no intervention. Those receiving the secure messaging program will receive an initial welcome message and monitoring messages approximately 2, 6, and 10 weeks after treatment has begun. The monitoring messages will include structured assessments of depression severity, medication adherence, medication side effects, and barriers to continuing treatment. Participants who do not respond to monitoring messages will receive up to two e-mailed reminders. Care managers will analyze the results of monitoring messages, provide feedback and recommendations to physicians, coordinate physician follow-ups, and facilitate emergency care or specialty referrals. Care managers will also provide patients with motivation, based on semi-scripted protocols, and education concerning their disorder and treatment. Measures of the success of the study will be taken at enrollment and after 6 months of participation. Specific measurements will include the response rate of recruitment e-mails, response rate for follow-up data collection, proportion of those in the secure messaging program who complete the monitoring assessments, effects of the program on antidepressant treatment, and effects of the program on patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Capitol Hill or Rainier clinics of Group Health Cooperative in Seattle
* New prescription of an antidepressant, defined by an interval of at least 180 days since a previous antidepressant prescription
* Indication of depression, defined by a visit diagnosis of major depressive disorder (Internal Classification of Diseases 9th Revision [ICD9] codes 296.2x or 296.3x) within 30 days of the first prescription
* Has used secure messaging, or e-mailing, at least twice in the last 12 months

Exclusion Criteria:

* Any diagnosis of psychotic disorder or bipolar disorder in the prior 2 years
* Any prescription for mood stabilizer or antipsychotic medication in the prior 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory E. Simon, MD, MPH, Principal Investigator — Group Health Cooperative Center for Health Studies
Locations (1):
- Group Health Cooperative Center for Health Studies, Seattle, Washington, United States

REFERENCES:
- [Result] Simon GE, Ralston JD, Savarino J, Pabiniak C, Wentzel C, Operskalski BH. Randomized trial of depression follow-up care by online messaging. J Gen Intern Med. 2011 Jul;26(7):698-704. doi: 10.1007/s11606-011-1679-8. Epub 2011 Mar 8. PMID 21384219

RESULTS

PARTICIPANT FLOW:
Groups:
- Secure Messaging Care Management: Participants will receive depression care management by secure messaging.
- Usual Care: Participants will receive their usual care, with no additional education or care management services.
Period: Overall Study
Arm/Group | Secure Messaging Care Management | Usual Care
Started | 106 | 102
Completed | 104 | 93
Not Completed | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secure Messaging Care Management | Usual Care | Total
Number analyzed (Participants) | 106 | 102 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 94 | 190
  >=65 years | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9) | 48 (10) | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 74 | 150
  Male | 30 | 28 | 58
Region of Enrollment [Number; unit: participants]
  United States | 106 | 102 | 208

OUTCOME MEASURES:

1. Primary Outcome: 20-Item Symptom Checklist Depression Scale
Description: 20-item depression severity scalse adapted from longer SCL-90. Mean score ranges from 0 to 4 with scores above 1.5 indicating moderate depression.
Time Frame: Measured at baseline and after 6 months of treatment
Population: Analysis included all participants participating in outcome assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Secure Messaging Care Management | Usual Care
Number analyzed (Participants) | 104 | 93
units on a scale | 0.95 (0.71) | 1.17 (0.81)

2. Secondary Outcome: Treatment Satisfaction
Description: Single item seven point scale ranging from "very satisfied" to "very dissatisfied"
Time Frame: Measured after 6 months of treatment
Measure: Number; unit: participants
Arm/Group | Secure Messaging Care Management | Usual Care
Number analyzed (Participants) | 104 | 93
participants
  Very Satisfied | 56 | 31
  Less than very satisfied | 48 | 62

ADVERSE EVENTS:
Arm/Group | Secure Messaging Care Management | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/93
Other Adverse Events (participants affected / at risk) | 0/104 | 0/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secure Messaging Care Management (N=104) | Usual Care (N=93)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0

LIMITATIONS AND CAVEATS:
Findings apply only to patients who choose to communicate by online messaging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No